CLINICAL TRIAL: NCT02371057
Title: The Prevalence of Acromegaly in the Sleep Apnoea Clinic
Brief Title: Acromegaly & Sleep Apnoea
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ED13/10973
Record Dates: First submitted 2015-02-11; First posted 2015-02-25 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients under follow-up known to have sleep apnoea
- patients attending the sleep apnoea clinic for assessment: Patients who are attending clinic who have not yet been diagnosed.

SUMMARY:
Estimates of the prevalence of acromegaly, a condition resulting from excess growth hormone secretion, are as high as 1:1000. If detected late acromegaly increases the risk of joint destruction, heart disease, sleep apnoea, high blood pressure, diabetes, and polyps in the colon. To have a greater effect on long-term outcomes this disease needs to be detected early. By screening a 'high risk' population (sleep apnoea clinic) the investigators may be able to detect these patients earlier and prevent late complications of the disease. At LTHT the referral pathway for new referrals to the sleep apnoea clinic involves initial attendance to pick up a pulse oximeter to wear overnight to measure oxygen levels. These readings show approximately 1:4 patients displays evidence of significant obstructive sleep apnoea to warrant referral to the treatment group for continuous positive airway pressure (CPAP), weight management, and occasionally mandibular adjustment.

Patients attending the sleep apnoea clinic either as new referral or for review will be asked to participate in the proposed study. The study is cross-sectional in design incorporating two sub-populations within the sleep apnoea clinic. The first cohort comprises patients under follow-up known to have sleep apnoea, and the second cohort those patients prospectively attending the sleep apnoea clinic for assessment. If after an explanation of the study they agree to participate blood will be taken for assessment of IGF-I and they will be asked to complete a simple questionnaire.

The aim will to be to screen 1000 consecutive patients. The questionnaire will incorporate five simple questions to be completed with a 'yes' or 'no' answer. Where IGF-I levels are elevated patients will be investigated further for the possibility of acromegaly. The presence of biochemically proven acromegaly will be used to determine if the simple question has sufficient sensitivity to use as a screening tool.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 16 and above.
* Referred to the Sleep Apnoea Clinic for assessment of obstructive sleep apnoea
* Have capacity to given informed consent.

Exclusion Criteria:

* Patients under 16 years of age
* Not referred to the Sleep Apnoea Clinic
* Unable to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients attending the sleep apnoea clinic.
Sampling Method: Probability Sample
Enrollment: 653 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
The prevalence of acromegaly within patients referred to the sleep apnoea clinic. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom